CLINICAL TRIAL: NCT05031104
Title: Efficacy of the Articular Application of Low-energy Laser on Knee Joints as an Auxiliary Treatment for Polyarticular Juvenile Idiopathic Arthritis: A Dual-arm Randomized Clinical Trial
Brief Title: Low-energy Laser Applications in Patients With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0018/027
Record Dates: First submitted 2021-08-28; First posted 2021-09-01 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Juvenile Idiopathic Arthritis; Rheumatic Diseases; Chronic Knee Pain; Fatigue; Muscle Weakness; Polyarticular JCA
MeSH Terms: conditions — Arthritis, Juvenile; Rheumatic Diseases; Fatigue; Muscle Weakness | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A prospective, dual-arm, randomized controlled trial with a 6-month follow-up
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients in this group undergone a standard exercise program.
  Interventions: Other: Physical Exercise
- LLT group (Experimental): Patients in this group undergone a standard exercise program as the control group in addition to the LLT.
  Interventions: Other: Physical Exercise plus Low-energy Laser Therapy

INTERVENTIONS:
Other: Physical Exercise — The control group received a standard exercise program for 40 minutes, three times a week for three successive months. The program encompassed aerobic, weight-bearing, proprioceptive, flexibility, and strengthening exercises.
  Arms: Control group
Other: Physical Exercise plus Low-energy Laser Therapy — The LLT group received the same program in addition to the application of LLT on both knees, each session before exercises.
  Arms: LLT group

SUMMARY:
This study endeavored to evaluate the auxiliary effect of low-energy laser therapy (LLT) on pain, muscle performance, fatigue, and functional ability in children with juvenile idiopathic arthritis (JIA). Sixty patients with JIA were randomly allocated to the LLT group (n = 30, received LLT in addition to the standard exercise program) or the control group (n = 30, received standard exercise program only). Both groups were assessed for pain intensity, muscle performance, fatigue perception, and functional status.

DETAILED DESCRIPTION:
Sixty patients with JIA were recruited from the Physical Therapy Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, and the Pediatric Rheumatology Clinic, King Khalid Hospital, Al-Kharj, Saudi Arabia. The study included patients who had a confirmed diagnosis of Polyarticular JIA (according to the criteria set forth by the International League of Associations for Rheumatology), aged 8-16 years, identified being stable cases, and did not participate in a regular exercise program (in the past six months). Patients who had fixed deformities, a history of joint surgery, or whose radiological investigations revealed erosive changes of bone, ankylosing, or fractures were excluded.

Outcome measures

1. Pain intensity: measures through the Visual Analogue Scale
2. Muscle performance: represented by the peak concentric torque of the right and left quadriceps muscle and measured through an Isokinetic Dynamometer.
3. Fatigue perception: tested by the Pediatric Quality of Life Inventory Multidimensional Fatigue Scale (PedsQL-MFS)
4. Functional status: the functional status was quantified using the cross-cultural validated version of the Childhood Health Assessment Questionnaire (CHAQ).

Patients in the control and LLT group received a 40-minute exercise program, three times a week, for three months in succession. Patients in the LLT group additionally underwent an articular application of LLT on the knee joint, each session before exercises (eight points on each knee, 30 seconds irradiation for each point, with a total irradiation dose of eight minutes per session. The treatment was conducted by two experienced pediatric physical therapists.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of JIA
* Polyarticular onset of JIA with bilateral involvement of the knee joint
* Age between 8 and 16 years
* Stable conditions (i.e., receive stable doses of medications in the past three months)
* Not participating in a regular exercise program in the past six months

Exclusion Criteria:

* Fixed deformities
* History of joint surgery
* Ankylosing or fractures
* Bone destruction (erosive changes of the knee joint)

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 2 months
  Pain intensity was measured through the Pain Visual Analogue Scale. Each child was asked to indicate his/her perceived pain intensity (most commonly) along a horizontal line (0-10 cm), where 0 represents "no pain" and 10 represents "worst pain".
Muscle performance | 2 months
  Represented by the peak concentric torque of the quadriceps muscle. It was measured using an Isokinetic Dynamometer.
Fatigue perception | 2 months
  The extent of fatigue that patients generally perceive was assessed using the Pediatric Quality of Life Inventory Multidimensional Fatigue Scale. Eighteen items across 3 subscales were rated on a 5-point Likert scale (0 = NEVER a problem and 4 = ALWAYS a problem). Item scores were linearly transformed on a 0-100 scale. The total score is calculated as the sum of all item scores divided by the number of rated items. Lower scores represent higher levels of fatigue perception.

SECONDARY OUTCOMES:
Functional status | 2 months
  The patient's ability to perform normal daily activities was assessed through the cross-culture validated version of the Childhood Health Assessment Questionnaire (parents-proxy report)

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Cairo University / Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No